CLINICAL TRIAL: NCT06707480
Title: Expanded Access Program to Provide Access to Defencath® for Adult and Pediatric Patients Using a Catheter to Prevent Central Line-Associated Bloodstream Infections (CLABSIs)
Brief Title: Expanded Access Program for Patients At Risk for Catheter-related Infections Who Are Not Eligible for DefenCath® Clinical Trials
Status: Available | Type: Expanded Access
Sponsor: CorMedix (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP-CLABSI
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Catheter-related Bloodstream Infection
MeSH Terms: interventions — taurolidine; Heparin

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Taurolidine and Heparin — Catheter Lock Solution
  Other Names: DefenCath®

SUMMARY:
The EAP for DefenCath is designed to provide access to a broader population of adult and pediatric patients using catheters for various serious medical conditions. A key aspect of this EAP is its focus on individuals who, due to their unique clinical circumstances, are either ineligible for participation in ongoing clinical trials or do not meet the criteria outlined in the current approved FDA label for DefenCath.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients: Male or female patients ≥18 years of age at the time of eligibility assessment, who are able and willing to provide informed consent.
* If the patient is unable to provide consent due to health status or mental capacity, a legally authorized representative (LAR) must provide written informed consent. Should the patient regain capacity, they must reconsent using the same consent form.
* Pediatric Patients: Male or female patients under 18 years of age at the time of eligibility assessment, with informed consent provided by an LAR if the patient is too young to consent or assent; patients capable of understanding the program may provide assent or full consent as appropriate.
* Patients receiving treatment through a catheter for serious medical conditions, including but not limited to hematologic and oncologic disorders, tumor-lysis syndrome, HD, TPN, peritoneal dialysis, intractable peritonitis, sickle-cell anemia and others. The catheter must be a permanent line made of silicone or polyurethane, in place for at least 7 days prior to enrollment. The specific type of catheter, e.g., peritoneal, tunneled, port-a-caths (ports), or peripherally inserted central catheter (PICC), must be documented.
* Patients who are able and willing to be trained, or have a caregiver, parent, or guardian capable of being trained, on the proper instillation and aspiration of DefenCath.
* Patients who have a minimum of a 4-hour CLS dwelling time.
* If female and of childbearing potential, the patient must have a negative pregnancy test at the screening visit (i.e., the subject is not pregnant); not be lactating; and use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or hormonal contraceptive (oral, implant, ring, patch) for the duration of the program. (NOTE: The subject must have used the chosen method of birth control for at least 1 month/cycle prior to enrollment into the EAP).
* Male patients who are sexually active with a female partner of childbearing potential must agree to use male condoms with spermicide, even if the male patient has undergone a successful vasectomy (males with vasectomy can use condoms without spermicide), from Day 1 until at least 30 days after the last DefenCath CLS installation.
* Patients who agree to adhere to all program procedures and follow-up requirements.
* Patients must have received approval from Supplier or its designee following the submission of the Treating Physician's request.

Exclusion Criteria:

* Patients with visible evidence of compromised skin integrity present at the catheter exit site or catheter exit site infection.
* Patients with a temporary, non-tunneled catheter.
* Patients who are eligible to participate in the ongoing clinical trials with DefenCath.
* Patients who are eligible to use DefenCath as per country approved label.
* Patients that have received thrombolytic treatment (e.g., tissue-type plasminogen activator [tPA]-Cathflo), not as a part of the institution's standard of care for patency management, in the current catheter within 30 days of enrolment into the EAP.
* Patients with a clinically significant medical condition that, in the opinion of the Treating Physician, pose a high risk of adverse outcomes or could compromise their safety during the EAP.
* Patients using any type of antimicrobial-coated or heparin-coated catheter.
* Patients with documented chronic bleeding diathesis, active or recurrent bleeding within 1 month prior to randomization.
* Patients with a congenitally lethal condition, a life expectancy of less than 3 months as determined by the Treating Physician.
* Patients with documented history of an atrial thrombus or known hypercoagulable state.
* Patients with known allergies or absolute contraindications to citrate, taurolidine, or heparin or a history of heparin-induced thrombocytopenia.
* Patients, or their immediate family members, who are the Treating Physician, sub-investigator, research assistant, pharmacist, site coordinator, or any other personnel directly involved in the conduct of the access program at the program site.

Sex: All
Age Groups: Child, Adult, Older Adult